CLINICAL TRIAL: NCT05092412
Title: A First-line Multi-center, Single-arm Exploratory Study Using Low-dose Radiotherapy (LDRT) Combined With Durvalumab (MEDI4736), Etoposide, and Cisplatin/Carboplatin for Patients With Extensive-stage Small Cell Lung Cancer
Brief Title: Low-dose Radiotherapy Combined With Durvalumab, Chemotherapy(EP) in the Treatment of ES-SCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: You Lu (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, You Lu, Professor, Sichuan University
Organization: Sichuan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-20-20849
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Extensive-stage Small-cell Lung Cancer; Durvalumab
Keywords: ES-SCLC; Durva; LDRT
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Radiotherapy; durvalumab; Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Low-dose radiotherapy combined with durvalumab, etoposide, and cisplatin/carboplatin (Experimental)
  Interventions: Radiation: Low-dose radiotherapy; Drug: Durvalumab; Drug: Etoposide, and cisplatin/carboplatin

INTERVENTIONS:
Radiation: Low-dose radiotherapy — The LDRT deals with primary tumour in a 15 Gy of 5fractions over five days, starting from Day 1 in the first cycle.
Drug: Durvalumab — Durvalumab 1500 mg intravenous infusion, started to be used simultaneously with chemotherapy at week 0 and continued after chemotherapy.
Drug: Etoposide, and cisplatin/carboplatin — Starting from week 0, the dose of etoposide + carboplatin or cisplatin in the study will not exceed the dose for specific indications in the product instructions (etoposide [80 to 100mg/m2] via intravenous infusion and carboplatin [ The area under the curve (AUC) is 5-6] by intravenous infusion or cisplatin [75-80 mg/m2] by intravenous infusion), using up to 4 cycles. The choice of platinum drugs is at the discretion of the investigator.

SUMMARY:
The purpose of this study was to evaluate the efficacy of low-dose radiotherapy (LDRT) combined with durvalumab, etoposide, and cisplatin/carboplatin in the first-line treatment of extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
This study will enrol 30 subjects at 3 sites in China. Subjects who fulfil all the inclusion criteria and none of the exclusion criteria will be enrolled and receive treatment with Durvalumab and EP for 4 cycles. Durvalumab will be administered at a dose of 1500 mg every 3 weeks (Q3W) with first-line chemotherapy and will continue to be administered as monotherapy every 4 weeks(Q4W) post-chemotherapy until progressive disease. The LDRT deals with primary tumour in a 15 Gy of 5 fractions over five days, starting from Day 1 in the first cycle. Subjects will attend safety follow up 12 weeks ±14 days after last dose of Durvalumab. The primary endpoint is mPFS.

ELIGIBILITY:
Inclusion Criteria:

* At the time of screening, male or female participants were ≥18 years old.
* Before carrying out any research program related procedures (including screening evaluation), obtain written informed consent and any locally required authorization from the participant or his legal representative.
* Extensive-stage disease confirmed by histology or cytology (American Joint Committee on Cancer (8th edition) stage IV SCLC [any T, any N and M1a/b/c]), or due to multiple lung nodules with a wide range Or the size of the tumor/nodule is too large to be included in a tolerable radiotherapy plan for stage T3-4 disease.

Participants with brain metastases must be asymptomatic or stable with steroids and anticonvulsants for at least 1 month before study treatment. Participants with suspected brain metastases during screening should undergo brain CT/MRI before enrollment in the study.

* The participant must be considered suitable for platinum-based chemotherapy as the first-line treatment for extensive-stage small cell lung cancer. Chemotherapy must include either cisplatin or carboplatin, combined with etoposide.
* The participant must be considered suitable for thoracic radiotherapy as the first-line treatment for extensive-stage small cell lung cancer.
* Life expectancy on the first day of study treatment was ≥12 weeks.
* At the time of enrollment, the World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) physical status score was 0 or 1.
* Weight>30 kg.
* According to the requirements of RECIST1.1 guidelines, at least one lesion (never received radiotherapy before), accurately measured by computed tomography (CT) or magnetic resonance imaging (MRI) at baseline shows that its longest diameter is ≥10mm (except for lymph nodes, Its short axis must be ≥15 mm); and the lesion is suitable for repeated and accurate measurement.
* Have not been exposed to immune-mediated therapies in the past, including but not limited to other anti-PD-1, anti-PD-L1 and anti-programmed cell death ligand 2 (anti-PD-L2) antibodies, except for therapeutic anti-tumor vaccines.
* With sufficient organ and bone marrow function, it needs to be measured 28 days before receiving treatment, which is defined as follows:

Hemoglobin ≥9 g/dL. Absolute neutrophil count ≥ 1.5 × 109/L (granulocyte colony stimulating factor is not allowed during screening).

Platelet count ≥75 × 109/L. Serum bilirubin ≤1.5 × upper limit of normal (ULN). It is not applicable to participants diagnosed with Gilbert syndrome. These participants are allowed to enter into the group through consultation with the investigators.

For participants without liver metastasis: ALT and AST ≤2.5 × ULN. The ALT and AST of participants with liver metastases are ≤5 × ULN.

* Measured or calculated creatinine clearance rate: According to the Cockcroft-Gault formula (using actual body weight) or a 24-hour urine test, participants receiving cisplatin therapy >60mL/min, and participants receiving carboplatin therapy >45mL/min.
* The female participant has evidence of postmenopausal status, or the urine or serum pregnancy test result of the premenopausal female participant is negative. Women who stop menopause for 12 months without other medical reasons are considered menopausal. The specific requirements for age are as follows:

For female participants <50 years of age who had amenorrhea for 12 months or more after discontinuing exogenous hormone therapy and whose luteinizing hormone and follicle-stimulating hormone levels were in the postmenopausal range or who had undergone sterilization (bilateral oophorectomy or hysterectomy) were considered postmenopausal.

For female participants ≥50 years of age, if all exogenous hormone treatments are stopped and the menopause is 12 months or more, or radiotherapy-induced ovariectomy and the last menstruation occurred more than 1 year ago, or chemotherapy-induced menopause and the last menstruation is more than 1 year , Or have undergone surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy), who can be considered a postmenopausal woman.

Exclusion Criteria:

* Participate in the design and execution of the study (applicable to researchers and/or members of the research center).
* Have previously received the distribution of experimental drug (IP) in this study.
* Enroll in another clinical study at the same time, unless it is an observational (non-interventional) clinical study or the follow-up phase of an interventional study.
* Etoposide-platinum (carboplatin or cisplatin)-based chemotherapy is medically contraindicated.
* Have a history of chest radiotherapy or plan to undergo intensive chest radiotherapy before systemic treatment. Radiotherapy outside the chest (eg, bone metastases) for the purpose of palliative care is allowed, but it must be completed before the first administration of the study drug.
* Simultaneously carry out any chemotherapy, biological products or hormone therapy for cancer treatment. The use of hormone therapy for non-cancer related conditions (eg, hormone replacement therapy) is acceptable.
* Major surgery (defined by the investigator) within 28 days before the first IP administration. Note: Local surgery on isolated lesions for the purpose of palliative care is acceptable.
* History of allogeneic organ transplantation.
* Paraneoplastic syndromes (PNS) with autoimmune properties requiring systemic treatment (systemic steroids or immunosuppressive agents) or clinical symptoms suggesting that PNS is aggravated.
* Active or previously recorded autoimmune diseases or inflammatory diseases (including inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [except diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, Wegener syndrome [granulomatous vasculitis, Graves disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). For this standard, the following exceptions:

Participants with vitiligo or hair loss. Participants with hypothyroidism (eg after Hashimoto syndrome) and stable disease after receiving hormone replacement therapy.

Any chronic skin disease that does not require systemic treatment. Participants without active disease in the past 5 years can be included in the study after discussion with the investigators.

Participants with celiac disease who can be controlled by diet alone.

* Uncontrolled concurrent diseases, including but not limited to: persistent or active infections, interstitial lung disease, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina, arrhythmia, concomitant Severe chronic gastrointestinal disease with diarrhea, or psychiatric/social problem conditions that may limit compliance with research requirements, cause a significant increase in the risk of AEs, or affect the participant's ability to provide written informed consent.
* A history of another type of primary malignant tumor, except for the following conditions:

Malignant tumors that are treated for the purpose of curing, have no known active disease ≥5 years before the first administration of IP, and have a low potential for recurrence risk.

Adequately treated non-melanoma skin cancer or malignant freckle-like nevus without evidence of disease.

Carcinoma in situ with adequate treatment and no evidence of disease.

* History of leptomeningeal carcinoma.
* History of active primary immunodeficiency.
* Active infections, including tuberculosis (clinical evaluation, including clinical history, physical examination, imaging findings and tuberculosis examination in line with local clinical practice), hepatitis B (known positive for HBV surface antigen [HbsAg]), hepatitis C or human immunity Defective virus (HIV 1/2 antibody positive). Participants who have previously suffered from HBV infection or who have been cured (defined as the presence of hepatitis B core IgG antibodies and the absence of HBsAg) are eligible. Participants who are positive for HCV antibodies are only eligible if they are negative for HCV RNA polymerase chain reaction.
* Immunosuppressive drugs were being used when durvalumab was first administered; Or use of immunosuppressive drugs in the 14 days prior to initial use of durvalumab. There are exceptions to this criterion:

Intranasal, inhaled, topical steroid therapy or local injection of steroid drugs (eg, intra-articular injection).

Systemic corticosteroid therapy that does not exceed 10 mg of prednisone per day or its equivalent physiological dose.

Steroids used as pre-medication for allergic reactions (for example, medication before CT scan). Steroid pretherapy for chemotherapy is acceptable.

* Vaccine live attenuated vaccine within 30 days before the first dose of IP. Note: After enrollment, participants cannot receive live vaccines during IP treatment and within 30 days after the last dose of IP.
* Pregnant or lactating female participants, or male or female participants with reproductive potential who are unwilling to take effective birth control measures during screening to 90 days after the last dosing of durvalumab monotherapy.
* Known to have allergic or hypersensitivity reactions to duvalvumab, etoposide, carboplatin, cisplatin or any of its excipients.
* Have participated in the clinical research of durvalumab and/or other anti-tumor drugs in the past, regardless of the allocation of treatment groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 2 years
  The time from the date of first dosing of durvalumab to the first appearance of objective disease progression (according to RECIST1.1) or death from any cause (if it occurs before disease progression).

SECONDARY OUTCOMES:
median overall survival（mOS） | up to 2 years
  Time from the date of first dosing of durvalumab to death from any cause.
Objective response rate (ORR) | up to 2 years
  According to the evaluation criteria of RECIST1.1.
6-month progression-free survival rate / 12-month progression-free survival rate (PFS6/12) | 1 years
  The proportion of patients who are still alive and have no disease progression 6 months/12 months after the first dose of Durvalumab.

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Study Chair — West China Hospital; Yan Zhang, MD, Principal Investigator — West China Hospital; Yue Xie, MM, Study Director — Chongqing University Cancer Hospital; Shu Jie Li, MM, Principal Investigator — Chongqing University Cancer Hospital; Shun Dong Cang, MD, Study Director — Henan Provincial People's Hospital; Lu Lu Su, MD, Principal Investigator — Henan Provincial People's Hospital
Locations (3):
- China (3):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - West China Hospital Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puglisi M, Dolly S, Faria A, Myerson JS, Popat S, O'Brien ME. Treatment options for small cell lung cancer - do we have more choice? Br J Cancer. 2010 Feb 16;102(4):629-38. doi: 10.1038/sj.bjc.6605527. Epub 2010 Jan 26. PMID 20104223
- [Background] Peifer M, Fernandez-Cuesta L, Sos ML, George J, Seidel D, Kasper LH, Plenker D, Leenders F, Sun R, Zander T, Menon R, Koker M, Dahmen I, Muller C, Di Cerbo V, Schildhaus HU, Altmuller J, Baessmann I, Becker C, de Wilde B, Vandesompele J, Bohm D, Ansen S, Gabler F, Wilkening I, Heynck S, Heuckmann JM, Lu X, Carter SL, Cibulskis K, Banerji S, Getz G, Park KS, Rauh D, Grutter C, Fischer M, Pasqualucci L, Wright G, Wainer Z, Russell P, Petersen I, Chen Y, Stoelben E, Ludwig C, Schnabel P, Hoffmann H, Muley T, Brockmann M, Engel-Riedel W, Muscarella LA, Fazio VM, Groen H, Timens W, Sietsma H, Thunnissen E, Smit E, Heideman DA, Snijders PJ, Cappuzzo F, Ligorio C, Damiani S, Field J, Solberg S, Brustugun OT, Lund-Iversen M, Sanger J, Clement JH, Soltermann A, Moch H, Weder W, Solomon B, Soria JC, Validire P, Besse B, Brambilla E, Brambilla C, Lantuejoul S, Lorimier P, Schneider PM, Hallek M, Pao W, Meyerson M, Sage J, Shendure J, Schneider R, Buttner R, Wolf J, Nurnberg P, Perner S, Heukamp LC, Brindle PK, Haas S, Thomas RK. Integrative genome analyses identify key somatic driver mutations of small-cell lung cancer. Nat Genet. 2012 Oct;44(10):1104-10. doi: 10.1038/ng.2396. Epub 2012 Sep 2. PMID 22941188
- [Background] Pignon JP, Arriagada R, Ihde DC, Johnson DH, Perry MC, Souhami RL, Brodin O, Joss RA, Kies MS, Lebeau B, et al. A meta-analysis of thoracic radiotherapy for small-cell lung cancer. N Engl J Med. 1992 Dec 3;327(23):1618-24. doi: 10.1056/NEJM199212033272302. PMID 1331787
- [Background] Roth BJ, Johnson DH, Einhorn LH, Schacter LP, Cherng NC, Cohen HJ, Crawford J, Randolph JA, Goodlow JL, Broun GO, et al. Randomized study of cyclophosphamide, doxorubicin, and vincristine versus etoposide and cisplatin versus alternation of these two regimens in extensive small-cell lung cancer: a phase III trial of the Southeastern Cancer Study Group. J Clin Oncol. 1992 Feb;10(2):282-91. doi: 10.1200/JCO.1992.10.2.282. PMID 1310103
- [Background] Rossi A, Di Maio M, Chiodini P, Rudd RM, Okamoto H, Skarlos DV, Fruh M, Qian W, Tamura T, Samantas E, Shibata T, Perrone F, Gallo C, Gridelli C, Martelli O, Lee SM. Carboplatin- or cisplatin-based chemotherapy in first-line treatment of small-cell lung cancer: the COCIS meta-analysis of individual patient data. J Clin Oncol. 2012 May 10;30(14):1692-8. doi: 10.1200/JCO.2011.40.4905. Epub 2012 Apr 2. PMID 22473169
- [Background] Clark R, Ihde DC. Small-cell lung cancer: treatment progress and prospects. Oncology (Williston Park). 1998 May;12(5):647-58; discussion 661-3. PMID 9597676
- [Background] Slotman BJ, van Tinteren H, Praag JO, Knegjens JL, El Sharouni SY, Hatton M, Keijser A, Faivre-Finn C, Senan S. Use of thoracic radiotherapy for extensive stage small-cell lung cancer: a phase 3 randomised controlled trial. Lancet. 2015 Jan 3;385(9962):36-42. doi: 10.1016/S0140-6736(14)61085-0. Epub 2014 Sep 14. PMID 25230595
- [Background] Reck M, Luft A, Szczesna A, Havel L, Kim SW, Akerley W, Pietanza MC, Wu YL, Zielinski C, Thomas M, Felip E, Gold K, Horn L, Aerts J, Nakagawa K, Lorigan P, Pieters A, Kong Sanchez T, Fairchild J, Spigel D. Phase III Randomized Trial of Ipilimumab Plus Etoposide and Platinum Versus Placebo Plus Etoposide and Platinum in Extensive-Stage Small-Cell Lung Cancer. J Clin Oncol. 2016 Nov 1;34(31):3740-3748. doi: 10.1200/JCO.2016.67.6601. PMID 27458307
- [Background] Dunn GP, Old LJ, Schreiber RD. The three Es of cancer immunoediting. Annu Rev Immunol. 2004;22:329-60. doi: 10.1146/annurev.immunol.22.012703.104803. PMID 15032581
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231
- [Background] Paterson AM, Brown KE, Keir ME, Vanguri VK, Riella LV, Chandraker A, Sayegh MH, Blazar BR, Freeman GJ, Sharpe AH. The programmed death-1 ligand 1:B7-1 pathway restrains diabetogenic effector T cells in vivo. J Immunol. 2011 Aug 1;187(3):1097-105. doi: 10.4049/jimmunol.1003496. Epub 2011 Jun 22. PMID 21697456
- [Background] Stewart R, Morrow M, Hammond SA, Mulgrew K, Marcus D, Poon E, Watkins A, Mullins S, Chodorge M, Andrews J, Bannister D, Dick E, Crawford N, Parmentier J, Alimzhanov M, Babcook JS, Foltz IN, Buchanan A, Bedian V, Wilkinson RW, McCourt M. Identification and Characterization of MEDI4736, an Antagonistic Anti-PD-L1 Monoclonal Antibody. Cancer Immunol Res. 2015 Sep;3(9):1052-62. doi: 10.1158/2326-6066.CIR-14-0191. Epub 2015 May 5. PMID 25943534
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Okudaira K, Hokari R, Tsuzuki Y, Okada Y, Komoto S, Watanabe C, Kurihara C, Kawaguchi A, Nagao S, Azuma M, Yagita H, Miura S. Blockade of B7-H1 or B7-DC induces an anti-tumor effect in a mouse pancreatic cancer model. Int J Oncol. 2009 Oct;35(4):741-9. doi: 10.3892/ijo_00000387. PMID 19724910
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Zhang C, Wu S, Xue X, Li M, Qin X, Li W, Han W, Zhang Y. Anti-tumor immunotherapy by blockade of the PD-1/PD-L1 pathway with recombinant human PD-1-IgV. Cytotherapy. 2008;10(7):711-9. doi: 10.1080/14653240802320237. PMID 18841514
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Planchard D, Yokoi T, McCleod MJ, Fischer JR, Kim YC, Ballas M, Shi K, Soria JC. A Phase III Study of Durvalumab (MEDI4736) With or Without Tremelimumab for Previously Treated Patients With Advanced NSCLC: Rationale and Protocol Design of the ARCTIC Study. Clin Lung Cancer. 2016 May;17(3):232-236.e1. doi: 10.1016/j.cllc.2016.03.003. Epub 2016 Mar 17. PMID 27265743
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Sandhu SK, Schelman WR, Wilding G, Moreno V, Baird RD, Miranda S, Hylands L, Riisnaes R, Forster M, Omlin A, Kreischer N, Thway K, Gevensleben H, Sun L, Loughney J, Chatterjee M, Toniatti C, Carpenter CL, Iannone R, Kaye SB, de Bono JS, Wenham RM. The poly(ADP-ribose) polymerase inhibitor niraparib (MK4827) in BRCA mutation carriers and patients with sporadic cancer: a phase 1 dose-escalation trial. Lancet Oncol. 2013 Aug;14(9):882-92. doi: 10.1016/S1470-2045(13)70240-7. Epub 2013 Jun 28. PMID 23810788
- [Background] Pacheco JM, Byers LA. Temozolomide plus PARP Inhibition in Small-Cell Lung Cancer: Could Patient-Derived Xenografts Accelerate Discovery of Biomarker Candidates? Cancer Discov. 2019 Oct;9(10):1340-1342. doi: 10.1158/2159-8290.CD-19-0850. PMID 31575562
- [Background] Wang Z, Sun K, Xiao Y, Feng B, Mikule K, Ma X, Feng N, Vellano CP, Federico L, Marszalek JR, Mills GB, Hanke J, Ramaswamy S, Wang J. Niraparib activates interferon signaling and potentiates anti-PD-1 antibody efficacy in tumor models. Sci Rep. 2019 Feb 12;9(1):1853. doi: 10.1038/s41598-019-38534-6. PMID 30755715
- [Background] Sen T, Rodriguez BL, Chen L, Corte CMD, Morikawa N, Fujimoto J, Cristea S, Nguyen T, Diao L, Li L, Fan Y, Yang Y, Wang J, Glisson BS, Wistuba II, Sage J, Heymach JV, Gibbons DL, Byers LA. Targeting DNA Damage Response Promotes Antitumor Immunity through STING-Mediated T-cell Activation in Small Cell Lung Cancer. Cancer Discov. 2019 May;9(5):646-661. doi: 10.1158/2159-8290.CD-18-1020. Epub 2019 Feb 18. PMID 30777870
- [Background] Paz-Ares L, Dvorkin M, Chen Y, Reinmuth N, Hotta K, Trukhin D, Statsenko G, Hochmair MJ, Ozguroglu M, Ji JH, Voitko O, Poltoratskiy A, Ponce S, Verderame F, Havel L, Bondarenko I, Kazarnowicz A, Losonczy G, Conev NV, Armstrong J, Byrne N, Shire N, Jiang H, Goldman JW; CASPIAN investigators. Durvalumab plus platinum-etoposide versus platinum-etoposide in first-line treatment of extensive-stage small-cell lung cancer (CASPIAN): a randomised, controlled, open-label, phase 3 trial. Lancet. 2019 Nov 23;394(10212):1929-1939. doi: 10.1016/S0140-6736(19)32222-6. Epub 2019 Oct 4. PMID 31590988
- [Background] Thomas A, Vilimas R, Trindade C, Erwin-Cohen R, Roper N, Xi L, Krishnasamy V, Levy E, Mammen A, Nichols S, Chen Y, Velcheti V, Yin F, Szabo E, Pommier Y, Steinberg SM, Trepel JB, Raffeld M, Young HA, Khan J, Hewitt S, Lee JM. Durvalumab in Combination with Olaparib in Patients with Relapsed SCLC: Results from a Phase II Study. J Thorac Oncol. 2019 Aug;14(8):1447-1457. doi: 10.1016/j.jtho.2019.04.026. Epub 2019 May 4. PMID 31063862
- [Background] Narod SA, Foulkes WD. BRCA1 and BRCA2: 1994 and beyond. Nat Rev Cancer. 2004 Sep;4(9):665-76. doi: 10.1038/nrc1431. PMID 15343273
- [Background] Chan KY, Ozcelik H, Cheung AN, Ngan HY, Khoo US. Epigenetic factors controlling the BRCA1 and BRCA2 genes in sporadic ovarian cancer. Cancer Res. 2002 Jul 15;62(14):4151-6. PMID 12124354
- [Background] Virag L, Szabo C. The therapeutic potential of poly(ADP-ribose) polymerase inhibitors. Pharmacol Rev. 2002 Sep;54(3):375-429. doi: 10.1124/pr.54.3.375. PMID 12223530
- [Background] Nguewa PA, Fuertes MA, Valladares B, Alonso C, Perez JM. Poly(ADP-ribose) polymerases: homology, structural domains and functions. Novel therapeutical applications. Prog Biophys Mol Biol. 2005 May;88(1):143-72. doi: 10.1016/j.pbiomolbio.2004.01.001. PMID 15561303
- [Background] Nishino M, Jagannathan JP, Ramaiya NH, Van den Abbeele AD. Revised RECIST guideline version 1.1: What oncologists want to know and what radiologists need to know. AJR Am J Roentgenol. 2010 Aug;195(2):281-9. doi: 10.2214/AJR.09.4110. PMID 20651182
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20104223/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22941188/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/1331787/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/1310103/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22473169/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/9597676/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25230595/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27458307/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15032581/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18173375/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17629517/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18500231/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21697456/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25943534/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22658128/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15705911/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12218188/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/19724910/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22658127/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18841514/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25428503/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27265743/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23945592/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23810788/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31575562/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30755715/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30777870/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31590988/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31063862/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15343273/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12124354/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12223530/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15561303/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/20651182/